CLINICAL TRIAL: NCT00001048
Title: A Phase II Multicenter Study Comparing Antiretroviral Therapy Alone to Antiretroviral Therapy Plus Cytosine Arabinoside (Cytarabine; Ara-C) for the Treatment of Progressive Multifocal Leukoencephalopathy (PML) in Human Immunodeficiency Virus (HIV)-Infected Subjects
Brief Title: Comparison of Anti HIV Drugs Used Alone or in Combination With Cytosine Arabinoside to Treat Progressive Multifocal Leukoencephalopathy (PML) in HIV-Infected Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Bristol-Myers Squibb (Industry); Upjohn (Industry)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: ACTG 243; 11220 (Registry Identifier: DAIDS-ES)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections; Leukoencephalopathy, Progressive Multifocal
Keywords: Leukoencephalopathy, Progressive Multifocal; Infusions, Intravenous; Cytarabine; Zalcitabine; Didanosine; Drug Therapy, Combination; Granulocyte Colony-Stimulating Factor; Acquired Immunodeficiency Syndrome; Zidovudine; Injections, Spinal
MeSH Terms: conditions — HIV Infections; Leukoencephalopathy, Progressive Multifocal; Acquired Immunodeficiency Syndrome | interventions — Filgrastim; Cytarabine; Zidovudine; Zalcitabine; Didanosine

INTERVENTIONS:
Drug: Filgrastim
Drug: Cytarabine
Drug: Zidovudine
Drug: Zalcitabine
Drug: Didanosine

SUMMARY:
To compare the safety and efficacy of antiretroviral therapy (zidovudine plus either didanosine or dideoxycytidine) versus antiretroviral therapy plus intravenous cytarabine (Ara-C) versus antiretroviral therapy plus intrathecal Ara-C in the maintenance or improvement of neurological function over 6 months in HIV-infected individuals who have developed progressive multifocal leukoencephalopathy (PML). To compare the effect of these three treatment regimens on Karnofsky score and MRI studies.

The effectiveness of Ara-C in the treatment of PML, caused by a human DNA papovavirus (designated JC virus) infection, has not been determined, although the most encouraging results have occurred with intrathecal administration of the drug.

DETAILED DESCRIPTION:
The effectiveness of Ara-C in the treatment of PML, caused by a human DNA papovavirus (designated JC virus) infection, has not been determined, although the most encouraging results have occurred with intrathecal administration of the drug.

Patients are randomized to receive antiretroviral therapy alone (AZT plus ddI or ddC), antiretroviral therapy plus intravenous Ara-C, or antiretroviral therapy plus intrathecal Ara-C. All patients receive 24 weeks of antiretroviral therapy. Beginning at week 2, patients on the intravenous Ara-C arm receive daily infusions of Ara-C over 5 days, with cycles repeating every 21 days. Patients on the intrathecal Ara-C arm receive single administrations of Ara-C at weeks 2, 3, 4, 5, 6, 8, 10, 12, 16, 20, and 24. A brain biopsy confirmation or in situ hybridization will be required within 7 days after study entry. Patients are followed every 4 weeks.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Local intralesional chemotherapy for mucocutaneous Kaposi's sarcoma.
* Topical antifungals, clotrimazole, ketoconazole, fluconazole, and amphotericin B for treatment of mucosal and esophageal candidiasis.
* Foscarnet for newly developed CMV infection, only after discussion with the protocol chair.
* Prophylactic and maintenance therapy for other opportunistic infections, provided patients are considered clinically stable.
* No more than 1000 mg/day acyclovir for herpes simplex.
* Antibiotics for bacterial infections as clinically indicated.
* Antipyretics, analgesics, and antiemetics.

Concurrent Treatment:

Allowed:

* Local radiation therapy for mucocutaneous Kaposi's sarcoma.

Patients must have:

* HIV infection.
* Confirmed PML.
* No other current active opportunistic infections requiring systemic therapy.
* Life expectancy of at least 3 months.

NOTE:

* A durable power of attorney is recommended where severe neurologic or psychiatric impairment can be foreseen while the patient is on study.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Current active cryptococcal meningitis, cytomegaloviral encephalitis, toxoplasmosis encephalitis, CNS lymphoma, or neurosyphilis.

NOTE:

* Patients on maintenance therapy for cryptococcal meningitis or toxoplasmosis encephalitis that has been stable for 4 months are permitted.
* Conditions that seriously increase risk of a surgical procedure (e.g., coagulopathy, severe thrombocytopenia).
* Any other disease that would interfere with evaluation of the patient.
* Other life-threatening complications likely to cause death in < 3 months.

Concurrent Medication:

Excluded:

* Ganciclovir.
* Interferon.
* Systemic chemotherapy other than Ara-C (unless specifically allowed).
* Antiretroviral medications other than AZT, ddI, or ddC.

Patients with the following prior conditions are excluded:

History of allergy or intolerance to G-CSF.

Prior Medication:

Excluded:

* Any prior Ara-C.

Excluded within 14 days prior to study:

* Ganciclovir or foscarnet.
* Interferon.
* Antiretroviral medications other than AZT, ddI, or ddC.
* Experimental medications for treatment of PML.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90
Dates: Study Completion 1997-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hall C, Study Chair; Timpone J, Study Chair
Locations (9):
- United States (9):
  - University of Colorado Hospital CRS, Aurora, Colorado
  - Univ. of Miami AIDS CRS, Miami, Florida
  - Northwestern University CRS, Chicago, Illinois
  - Johns Hopkins Adult AIDS CRS, Baltimore, Maryland
  - Massachusetts General Hospital ACTG CRS, Boston, Massachusetts
  - Washington U CRS, St Louis, Missouri
  - Univ. of Rochester ACTG CRS, Rochester, New York
  - Unc Aids Crs, Chapel Hill, North Carolina
  - University of Washington AIDS CRS, Seattle, Washington

REFERENCES:
- [Background] Cytarabine nixed for PML. GMHC Treat Issues. 1996 Nov;10(11):9. PMID 11364014
- [Background] Post MJ, Yiannoutsos C, Simpson D, Booss J, Clifford DB, Cohen B, McArthur JC, Hall CD. Progressive multifocal leukoencephalopathy in AIDS: are there any MR findings useful to patient management and predictive of patient survival? AIDS Clinical Trials Group, 243 Team. AJNR Am J Neuroradiol. 1999 Nov-Dec;20(10):1896-906. PMID 10588116
- [Background] Hall C, Timpone J, Dafni I, Antonijevic Z, Millar L, Booss J, Clifford D, Cohen B, McArthur J, Hollander H. ARA-C treatment of PML in AIDS patients. Conf Retroviruses Opportunistic Infect.1997 Jan 22-26;4th:66 (abstract no 8)PMID: 97926517
- [Background] Yiannoutsos CT, Major EO, Curfman B, Jensen PN, Gravell M, Hou J, Clifford DB, Hall CD. Relation of JC virus DNA in the cerebrospinal fluid to survival in acquired immunodeficiency syndrome patients with biopsy-proven progressive multifocal leukoencephalopathy. Ann Neurol. 1999 Jun;45(6):816-21. doi: 10.1002/1531-8249(199906)45:63.0.co;2-w. PMID 10360779
- [Background] Hall CD, Dafni U, Simpson D, Clifford D, Wetherill PE, Cohen B, McArthur J, Hollander H, Yainnoutsos C, Major E, Millar L, Timpone J. Failure of cytarabine in progressive multifocal leukoencephalopathy associated with human immunodeficiency virus infection. AIDS Clinical Trials Group 243 Team. N Engl J Med. 1998 May 7;338(19):1345-51. doi: 10.1056/NEJM199805073381903. PMID 9571254
- [Background] Crit Path AIDS Proj 1994-95 Winer; (No 30): 28-29. A phase II Multicenter Study Comparing Antiretroviral Therapy Alone to Antiretroviral Therapy Plku Cytosine Arabinosine (Cytarabine; Ara-C) for the Treatment of Progressive Multifocal Leukoencephalopathy (PML) in Human Immunodeficiency Virus (HIV)-Infected Subjects. .